CLINICAL TRIAL: NCT02462655
Title: Effects of LDL Apheresis System on the Expression of Genes Involved in Lipoprotein Metabolism and Inflammation in Homozygotes for Familial Hypercholesterolemia
Acronym: LA-PBMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Patrick Couture, MD, PHD, FRCP, Laval University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LA-PBMC
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-lipid apheresis (Experimental): Blood samples will be taken just before the start of the lipid apheresis treatment.
  Interventions: Other: Pre-lipid apheresis
- Post-lipid apheresis (Experimental): Blood samples will be taken following the lipid apheresis treatment.
  Interventions: Other: Post-lipid apheresis

INTERVENTIONS:
Other: Pre-lipid apheresis — Blood samples will be taken just before the start of the lipid apheresis treatment.
  Arms: Pre-lipid apheresis
Other: Post-lipid apheresis — Blood samples will be taken following the lipid apheresis treatment.
  Arms: Post-lipid apheresis

SUMMARY:
Familial hypercholesterolemia (FH) is an autosomal codominant single-gene disorder caused by mutations in the LDL receptor gene that disrupt the normal clearance of LDL particles from the plasma compartment. Heterozygous patients present a 2- to 3-fold raise in plasma LDL-cholesterol (C) concentrations, tendinous xanthomatosis and premature atherosclerotic coronary heart disease (CHD), usually occurring between the age of 35 and 55 years. Since the mid-1970s, LDL-C has been removed from the blood of patients using plasmapheresis, and this technique has been shown to improve the life expectancy of FH homozygotes. LDL apheresis selectively removes LDL particles but not immunoglobulins and other beneficial proteins, thereby overcoming a potential drawback of the traditional plasmapheresis method. LDL-C is effectively reduced by more than 60% immediately after LDL apheresis, although LDL levels rebound rapidly.

Dextran sulfate adsorption is a commonly apheresis technique used in familial hypercholesterolemia patients. In this apheresis plasma is separated from red blood cells and passed over columns of cellulose beads containing dextran sulfate which binds apolipoprotein B (apoB) by a highly selective electrostatic binding mechanism. Since LDL, very-low density lipoprotein (VLDL), and Lipoprotein (a) all contain apoB, dextran sulfate adsorption apheresis selectively reduces these lipoproteins while having little effect on the non-apoB containing HDL particles. In clinical practice, LDL apheresis reduces the rate of future cardiovascular events and has been postulated to have additional effects on potentially pro-atherogenic factors. Some proteins have been identified with adhesive characteristics to lipoproteins, rheological, immunological and inflammation relevant proteins16-19 that influence microcirculation as well as the inflammatory response. However, no studies have yet to investigate the impact of LDL apheresis on the expression of different genes involved in cardiovascular disease.

The main objective of the present research project is to investigate the impact of the LDL apheresis dextran sulfate adsorption system on the messenger ribonucleic acid (mRNA) expression of genes involved in cardiovascular disease using microarrays analysis in 9 FH homozygotes.

ELIGIBILITY:
Inclusion Criteria:

* Homozygotes for familial hypercholesterolemia who receive lipid apheresis
* Aged between 18-60 years

Exclusion Criteria:

* Smokers (> 1 cigarette/day)
* Subjects with a previous history of cardiovascular disease
* Subjects with type 2 diabetes
* Subjects with a monogenic dyslipidemia that it is not homozygote for familial hypercholesterolemia
* Subjects with endocrine or gastrointestinal disorders
* History of alcohol or drug abuse within the past 2 years
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in mRNA expression of genes involved in cardiovascular disease using microarrays analysis. | Pre-lipid apheresis (t=0h) and post-lipid apheresis (t=3h)

SECONDARY OUTCOMES:
Change in serum levels of C-reactive protein | Pre-lipid apheresis (t=0h) and post-lipid apheresis (t=3h)

OTHER OUTCOMES:
Change in serum levels of vascular cell adhesion molecule | Pre-lipid apheresis (t=0h) and post-lipid apheresis (t=3h)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD,FRCP,PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Québec, Quebec, Canada